CLINICAL TRIAL: NCT00425152
Title: A Clinical Trial to Assess the Relative Efficacy of 5-FU + Leucovorin, 5-FU + Levamisole, and 5-FU + Leucovorin + Levamisole in Patients With Dukes' B and C Carcinoma of the Colon
Brief Title: Fluorouracil and Leucovorin and/or Levamisole After Surgery In Treating Patients With Dukes' B Or Dukes' C Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Northern California Cancer Center (Other)
Responsible Party: Norman Wolmark, MD, NSABP Foundation, Inc.
Purpose: Treatment
Other Study IDs: NSABP C-04; U10CA012027 (NIH); NCOG-NSABP-C-04
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Leucovorin; Levamisole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: levamisole hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Leucovorin may help fluorouracil kill more tumor cells. Biological therapies, such as levamisole, may interfere with the growth of tumor cells and slow the growth of solid tumors. It is not yet known whether fluorouracil is more effective when given together with leucovorin and/or levamisole after surgery in treating colon cancer.

PURPOSE: This randomized phase III trial is studying giving fluorouracil together with leucovorin to see how well it works compared with giving fluorouracil together with levamisole, or giving fluorouracil together with leucovorin and levamisole after surgery in treating patients with Dukes' B or Dukes' C colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare, in a Phase III setting, disease-free survival and overall survival of patients who have undergone potentially curative resection of Dukes' B or C carcinoma of the colon randomly assigned to adjuvant therapy with 5-fluorouracil/leucovorin vs. 5-fluorouracil/levamisole vs. 5-fluorouracil/leucovorin/levamisole.

OUTLINE: Randomized study. Arm I: Single-agent Chemotherapy with Drug Modulation. 5-Fluorouracil, 5-FU, NSC-19893; with Leucovorin calcium, Citrovorum Factor, CF, NSC-3590. Arm II: Single-agent Chemotherapy with Drug Modulation plus Biological Response Modifier Therapy. 5-FU; with CF; plus Levamisole, LEV, NSC-177023. Arm III: Single-agent Chemotherapy plus Biological Response Modifier Therapy. 5-FU; plus LEV.

PROJECTED ACCRUAL: 1,800 evaluable patients will be accrued over about 3 years; an additional 2 years will be required before final analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: See General Eligibility Criteria

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2151 (Actual)
Dates: Start 1989-07; Primary Completion 1998-06 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Study Chair — Allegheny Cancer Center at Allegheny General Hospital; Robert W. Carlson, MD, Study Chair — Stanford University

REFERENCES:
- [Background] Wilkinson NW, Yothers G, Lopa SH, et al.: Long-term survival results of surgery alone compared with surgery plus 5-fluorouracil and leucovorin for stage II and stage III colon cancer: pooled analysis of NSABP adjuvant trials C-01 through C-05. [Abstract] American Society of Clinical Oncology 2009 Gastrointestinal Cancers Symposium, 15-17 January 2009, San Francisco, CA. A-442, 2009.
- [Background] Kim GP, Colangelo LH, Wieand HS, Paik S, Kirsch IR, Wolmark N, Allegra CJ; National Cancer Institute. Prognostic and predictive roles of high-degree microsatellite instability in colon cancer: a National Cancer Institute-National Surgical Adjuvant Breast and Bowel Project Collaborative Study. J Clin Oncol. 2007 Mar 1;25(7):767-72. doi: 10.1200/JCO.2006.05.8172. Epub 2007 Jan 16. PMID 17228023
- [Background] Dignam JJ, Polite BN, Yothers G, Raich P, Colangelo L, O'Connell MJ, Wolmark N. Body mass index and outcomes in patients who receive adjuvant chemotherapy for colon cancer. J Natl Cancer Inst. 2006 Nov 15;98(22):1647-54. doi: 10.1093/jnci/djj442. PMID 17105987
- [Background] Wang SJ, Zamboni BA, Wieand HS, et al.: Conditional survival for patients with colon cancer: an analysis of National Surgical Adjuvant Breast and Bowel Project (NSABP) trials C-03 through C-06. [Abstract] J Clin Oncol 24 (Suppl 18): A-6005, 302s, 2006.
- [Background] Allegra CJ, Paik S, Colangelo LH, Parr AL, Kirsch I, Kim G, Klein P, Johnston PG, Wolmark N, Wieand HS. Prognostic value of thymidylate synthase, Ki-67, and p53 in patients with Dukes' B and C colon cancer: a National Cancer Institute-National Surgical Adjuvant Breast and Bowel Project collaborative study. J Clin Oncol. 2003 Jan 15;21(2):241-50. doi: 10.1200/JCO.2003.05.044. PMID 12525515
- [Background] Wolmark N, Colangelo L, Wieand S. National Surgical Adjuvant Breast and Bowel Project trials in colon cancer. Semin Oncol. 2001 Feb;28(1 Suppl 1):9-13. doi: 10.1016/s0093-7754(01)90245-3. PMID 11273592
- [Background] Dignam JJ, Colangelo L, Tian W, Jones J, Smith R, Wickerham DL, Wolmark N. Outcomes among African-Americans and Caucasians in colon cancer adjuvant therapy trials: findings from the National Surgical Adjuvant Breast and Bowel Project. J Natl Cancer Inst. 1999 Nov 17;91(22):1933-40. doi: 10.1093/jnci/91.22.1933. PMID 10564677
- [Background] Mamounas E, Wieand S, Wolmark N, Bear HD, Atkins JN, Song K, Jones J, Rockette H. Comparative efficacy of adjuvant chemotherapy in patients with Dukes' B versus Dukes' C colon cancer: results from four National Surgical Adjuvant Breast and Bowel Project adjuvant studies (C-01, C-02, C-03, and C-04). J Clin Oncol. 1999 May;17(5):1349-55. doi: 10.1200/JCO.1999.17.5.1349. PMID 10334518
- [Result] Wolmark N, Rockette H, Mamounas E, Jones J, Wieand S, Wickerham DL, Bear HD, Atkins JN, Dimitrov NV, Glass AG, Fisher ER, Fisher B. Clinical trial to assess the relative efficacy of fluorouracil and leucovorin, fluorouracil and levamisole, and fluorouracil, leucovorin, and levamisole in patients with Dukes' B and C carcinoma of the colon: results from National Surgical Adjuvant Breast and Bowel Project C-04. J Clin Oncol. 1999 Nov;17(11):3553-9. doi: 10.1200/JCO.1999.17.11.3553. PMID 10550154
- [Result] Wolmark N, Rockette H, Mamounas EP, et al.: The relative efficacy of 5-FU + leucovorin (FU-LV), 5-FU + levamisole (FU-LEV), and 5-FU + leucovorin + levamisole (FU-LV-LEV) in patients with Dukes' B and C carcinoma of the colon: first report of NSABP C-04. [Abstract] Proceedings of the American Society of Clinical Oncology 15: A460, 205a, 1996.
- [Derived] Yothers G, Sargent DJ, Wolmark N, Goldberg RM, O'Connell MJ, Benedetti JK, Saltz LB, Dignam JJ, Blackstock AW; ACCENT Collaborative Group. Outcomes among black patients with stage II and III colon cancer receiving chemotherapy: an analysis of ACCENT adjuvant trials. J Natl Cancer Inst. 2011 Oct 19;103(20):1498-506. doi: 10.1093/jnci/djr310. Epub 2011 Oct 12. PMID 21997132